CLINICAL TRIAL: NCT06062498
Title: Randomized Phase II Study of Elacestrant vs Elacestrant Plus a CDK4/6 Inhibitor (Palbociclib, Abemaciclib, or Ribociclib) in Patients With ER+/HER2- Advanced or Metastatic Breast Cancer With Prior Exposure to a CKD4/6 Inhibitor
Brief Title: Elacestrant vs Elacestrant Plus a CDK4/6 Inhibitor in Patients With ERpositive/HER2-negative Advanced or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 23B05; STU00219978 (Other: NU IRB); NU 23B05 (Other: Northwestern University); NCI-2023-07168 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA060553 (NIH)
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Estrogen-receptor-positive Breast Cancer; HER2/Neu-Negative Breast Cancer; Advanced Breast Cancerv; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; palbociclib; abemaciclib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elacestrant Monotherapy (Experimental): Elacestrant (345 mg) will be taken orally once daily for each 28-day cycle. Courses repeat until progressive disease.
  Interventions: Drug: elacestrant, palbociclib, abemaciclib, ribociclib
- Combination Therapy (Experimental): Patients will receive either:
  Elacestrant 345 mg orally once daily
  + Palbociclib 125 mg orally once daily for 21 days out of 28-day cycle OR Abemaciclib 150 mg orally twice daily OR Ribociclib 600 mg orally once daily for 21 days out of 28-day cycle
  Interventions: Drug: elacestrant, palbociclib, abemaciclib, ribociclib

INTERVENTIONS:
Drug: elacestrant, palbociclib, abemaciclib, ribociclib — Given orally

SUMMARY:
Breast cancer is not only the leading cause of cancer in women, but also the leading cause of cancer deaths in women. Estrogen receptor-positive and HER2-negative breast cancer is the most prevalent breast cancer subtype. Endocrine therapy is the mainstay of treatment; however, due to the varied nature of the disease, development of resistance to this therapeutic approach is very common in the metastatic setting.

The purpose of this study is to see whether the effectiveness of elacestrant can be enhanced by combining it with a targeted agent such as a CDK4/6 inhibitor to treat patients with ER+/HER2- or metastatic breast cancer with prior exposure to a CDK4/6 inhibitor.

DETAILED DESCRIPTION:
Primary Objective I. Evaluate progression-free survival (PFS) of patients with advanced or metastatic ERpositive/HER2-negative breast cancer who have been treated with either elacestrant monotherapy or combination therapy of elacestrant with a CDK4/6 inhibitor (palbociclib, abemaciclib, or ribociclib). PFS of the elacestrant monotherapy arm will be compared with PFS of the combination therapy arm.

Secondary Objectives I. Assess toxicity profile of elacestrant combination therapy with a CDK4/6 inhibitor (palbociclib, abemaciclib, or ribociclib) in advanced or metastatic ER-positive/HER2- negative breast cancer according to NCI-CTCAE v5.0.

II. Assess duration of response (DOR) in patients with advanced or metastatic ERpositive/HER2-negative breast cancer who have been treated with either elacestrant monotherapy or combination therapy of elacestrant with a CDK4/6 inhibitor (palbociclib, abemaciclib, or ribociclib). DOR of the elacestrant monotherapy arm will be compared with DOR of the combination therapy arm. III. Determine overall survival (OS) in patients with advanced or metastatic ER-positive, HER2-negative breast cancer who have been treated with either elacestrant monotherapy or combination therapy of elacestrant with a CDK4/6 inhibitor (palbociclib, abemaciclib, or ribociclib). OS of the elacestrant monotherapy arm will be compared with OS of the combination therapy arm.

OUTLINE:

Patients will receive either elacestrant monotherapy or combination therapy with a CDK4/6 inhibitor (palbociclib, abemaciclib, or ribociclib) orally for each 28 day cycle until progressive disease, unacceptable toxicity, treating physician decision, or patient withdrawal of consent.

Patients will be followed (either by routine clinic visit or by phone call) every 36 weeks for 2 years and then every 72 weeks up to 5 years total from time of registration to document survival and disease progression.

ELIGIBILITY:
Inclusion Criteria All Arms:

* Patients must have histologically or cytologically confirmed ER-positive and HER2- negative breast cancer as per the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines (Allison et al, 2020, Wolff et al, 2018).

Note: In the context of this trial, ER status will be considered positive if >10% of tumor cells demonstrate positive nuclear staining by immunohistochemistry. Note: Fresh biopsy is not a requirement.

* Patients must have a confirmed ESR1 mutation. Note: This information will be drawn from patients' treatment charts. Mutational analysis will be done as standard of care; there is no research-related mutational testing for this study. ctDNA may be used for mutational testing.
* Patients must have at least one measurable lesion (as per RECIST v1.1) lesion anywhere in the body or a mainly lytic metastatic bone lesion. Note: Lytic bone lesions with identifiable soft tissue components that can be evaluated by cross-sectional imaging techniques such as CT or MRI can be considered as measurable lesions if the soft tissue component meets the definition of measurability per RECIST v1.1.
* Patients must have received at least 2 prior endocrine therapies, including a CDK4/6 inhibitor in the metastatic disease setting.
* Patients must be age ≥ 18 years. Patients of childbearing potential (POCBP) may be premenopausal, postmenopausal, or perimenopausal.
* Potential POCBP who may be menopausal and are < 55 years of age must have a serum follicle-stimulating hormone (FSH) level > 40 mIU/mL to confirm menopause.
* Patients must exhibit an ECOG performance status of 0 or 1.
* Patients must have adequate organ and bone marrow function as defined below:

Leukocytes (WBC) ≥ 3,000/mcL Absolute neutrophil count (ANC) ≥ 1,500/mcL Hemoglobin (Hgb) ≥ 80-100 g/dL Platelets (PLT) ≥ 50,000/mcL Total serum bilirubin < 1.5 x Institutional upper limit of normal (ULN) AST (SGOT) ≤ 3 x institutional ULN (no liver metastases)

* 5 x institutional ULN (liver metastases present) ALT (SGPT) ≤ 3 x institutional ULN
* 5 x institutional ULN (liver metastases present) Cockcroft-Gault based creatinine clearance

  * 50 mL/min

Note:

* Creatinine clearance (DMAB)

  = ([140-age in years] × weight in kg)/ ([serum creatinine in mg/dL] × 72)
* Creatinine clearance (DFAB) = (0.85 × [140-age in years] × weight in kg)/ ([serum creatinine in mg/dL] × 72) Note: Growth factor/transfusion support to attain these levels is not permitted.

  * For patients with a known history of human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy must have a viral load undetectable for 6 months prior to registration.
  * For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
  * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are eligible.
  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better. Elacestrant is a known teratogen. For this reason, patients of child-bearing potential (POCBP) and their partners with sperm-producing reproductive capacity must agree to use adequate contraception (see Appendix B) from time of informed consent, for the duration of study participation, and for 7 days following completion of elacestrant therapy.

Should a POCBP become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately. Patients with sperm-producing reproductive capacity (PWSPRC) treated or enrolled on this protocol must also agree to use adequate contraception with partners of childbearing potential from time of informed consent, for the duration of study participation, and 7 days after completion of administration. Note: A POCBP is any patient (regardless of gender, sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) with an egg-producing reproductive tract who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months) Note: POCBP who are on combination therapy with any study CKD4/6 inhibitor (palbociclib, abemaciclib, or ribociclib) must agree to use adequate contraception from time of informed consent, for the duration of study participation, and for 21 days following completion of CKD4/6 inhibitor therapy. POCBP must have a negative pregnancy test prior to registration on study. If initial urine pregnancy test is positive or cannot be confirmed negative, serum pregnancy test will be required. -Patients must have the ability to understand and the willingness to sign a written informed consent document.

Inclusion Criteria - Combination Therapy Arm 2 with Palbociclib, Abemaciclib, or Ribociclib

-Patients who have been treated with one or two prior hormonal therapies in the metastatic setting if at least one hormonal therapy was in combination with a CDK4/6 inhibitor.

Notes:

* Patients who are already on or have already been exposed to one or two of the study CDK4/6 inhibitors at registration will be assigned a different study CDK4/6 inhibitor (e.g., if a patient has already been exposed to abemaciclib, they will be given ribociclib or palbociclib; similarly, if a patient has already been exposed to palbociclib and abemaciclib, they will be given ribociclib.)
* One-to-one randomization will be done by the QA team once patients have been registered.

Exclusion Criteria All Arms:

* Patients who have received prior elacestrant.
* Patients who have had chemotherapy or radiotherapy ≤ 28 days (6 weeks for nitrosureas or mitomycin C) prior to registration.
* Patients who have taken steroid therapy or any other immunosuppressive therapy within 7 days of first dose prior to trial treatment.
* Patients with brain metastases. Note: Patients with stable brain or subdural metastases are allowed if the patient has completed local therapy and was on a stable or decreasing dose of corticosteroids at baseline for brain management for at least 4 weeks before starting treatment in this study. The dose must be <2.0 mg/day of dexamethasone or equivalent. Any signs (e.g., radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment. RANO criteria are used to evaluate brain metastases
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 3) with the exception of alopecia.
* Patients who are receiving any other investigational agents. For patients who were previously on palbociclib, abemaciclib, or ribociclib, the washout period between stopping that CDK4/6 inhibitor and starting a different one is 14 days.
* Patients with advanced, symptomatic visceral spread who are at risk of life-threatening complications in the short term, including massive uncontrolled effusions (peritoneal, pleural, pericardial), pulmonary lymphangitis, or liver involvement >50%.
* Patients with documented pneumonitis/interstitial lung disease prior to registration.
* Patients who have received major surgery within 28 days before starting trial therapy.
* Patients who are taking strong or moderate CYP3A4 inducers or strong or moderate CYP3A4 inhibitors. See Section 4.4 for additional incompatibilities.
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to elacestrant. Note: Refer to exclusion criteria below for eligibility criteria related to study CDK4/6 inhibitors.
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Hypertension that is not controlled on medication
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients with refractory or chronic nausea, gastrointestinal conditions (including significant gastric or bowel resection or gastric bypass surgery), history of malabsorption syndrome, or any other uncontrolled gastrointestinal condition that impact the absorption of the study drug. Similarly, patients who are unable to take/retain oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years
  The primary endpoint of PFS for elacestrant or combination therapy (elacestrant and either palbociclib, abemaciclib, or ribociclib) will involve calculation of the progression-free survival time as the time that elapses between time of treatment initiation and first documented disease progression or death from any cause (whichever comes first). For PFS analysis, disease progression is defined as progressive disease (PD) per RECIST v1.1. The PFS results from the two treatment arms will be compared.

SECONDARY OUTCOMES:
Adverse events | Up to 30 business days after end of treatment
  To determine toxicity, grading will be evaluated using NCI CTCAE v5.0. Adverse events will be assessed from start of therapy up to 30 business days after treatment discontinuation.
Duration of Response (DOR) | Up to 5 years
  For DOR analysis, response is defined as confirmed complete response (CR) or confirmed partial response (PR) per RECIST v1.1. Disease progression is defined as progressive disease (PD) per RECIST v1.1.
Overall Survival (OS) | Up to 5 years
  Overall survival is calculated as the time that elapses between the day of patient registration and death from any cause, for all evaluable patients.

CONTACTS AND LOCATIONS:
Overall Officials: William Gradishar, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No